CLINICAL TRIAL: NCT07343713
Title: Correlation Between the Degree of Middle Ear Pressure and the Eustachian Tube Dimensions : Radiological Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khloud youssef sayed abdallah, Postgraduate Researcher, Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: khloud youssef sayed abdallah
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: the Degree of Middle Ear Pressure and the Eustachian Tube Dimensions
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — No intervention was applied. This is an observational study in which participants underwent routine clinical and radiological assessments only, with no experimental or therapeutic intervention.

SUMMARY:
The eustachian tube (ET) as it is known has important tasks on middle ear function and physiology. Middle ear ventilation, drainage, and protection of the middle ear to pathogens are major functions of the eustachian tube. Earlier studies showed that the eustachian tubes were shorter and were more horizontally located in children than in adults. This condition might increase otitis media in children (1).

The angles relative to the plane of the eustachian tube have previously been measured in a lot of work. These measurements were obtained in mostly cadaver studies. In various studies with the temporal bone computed tomography (CT), the eustachian tube placement was assessed according to the relationship to other structures (2).

Reid horizontal plane was found in 1962 by the world federation of radiology, bilateral inferior orbital wall and superior walls of the bilateral external ear canal. This plane is considered to be the position at which the head in a neutral anatomical position. Reid plane of eustachian tube angle is defined as the angle between tympanic pharyngeal orifice and Reid plane. Tubotympanic angle is an angle more recently associated with COM and cholesteatoma.This angle is defined as the angle of the longitudinal axis of the eustachian tube along the tympanic orifice and the longitudinal axis of the center the bony external ear canal of the bone in the axial plane(3).

There was a positive correlation between the degree of the mastoid pneumatization and the eustachian tube length (4). The decrease in the angle with the horizontal plane of Reid in the Eustachian tube in adults may play a significant role in the etiology of cholesteatoma(1).

ELIGIBILITY:
Inclusion Criteria:

* healthy tympanic membrane age more than 7 years

Exclusion Criteria:

* i. Childern before 7 years. ii. Unhealthy tympanic membrane. iii. Patients with any kind of otitis media. iv. Patients with upper respiratory tract infection. v. Previous radiotherapy. vi. Patients with gastroesophageal reflux. vii. Previous temporal bone trauma.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 7-18 years attending the ENT clinic at Assiut University Children's Hospital, with no prior ear surgery or chronic ear disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical and functional parameters of the Eustachian tube | Single assessment at the time of imaging or clinical evaluation

IPD SHARING:
Plan to Share IPD: No